CLINICAL TRIAL: NCT02717741
Title: A Phase I Study to Determine the Safety and Pharmacokinetic Study of Tafetinib in Patients With Advanced Solid Tumors
Brief Title: A Study of Tafetinib in Chinese Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NanjingYoko
Record Dates: First submitted 2016-03-03; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — N-(2-(diethylamino)ethyl)-2-methyl-7-(1,2-dihydro-5-fluoro-2-oxo-3H-indol-3-ylidene)-4,5,6,7-tetrahydro-1H-indole-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tafetinib (Experimental): tafetinib administered daily for 2 weeks, followed by a 1-week off period
  Interventions: Drug: tafetinib

INTERVENTIONS:
Drug: tafetinib

SUMMARY:
Tafetinib is an oral multitargeted tyrosine kinase inhibitor that inhibits Vascular Endothelial Growth Factor Receptor (VEGFR).

This phase I trial was conducted to evaluate the pharmacokinetics (PK), safety, and preliminary efficacy of tafetinib in Chinese patients with advance solid tumor. The study are conducting in Cancer Hospital Chinese Academy of Medical Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically confirmed advanced solid malignancies.
* ECOG score 0-1.
* 18-65 years old.
* Withdrawal other chemotherapy drugs more than 30 days. No nitrosoureas or mitomycin C within the previous 6 weeks.
* Function of organs must meet the following requirements:
* Neutrophil count ≥1500/ul;
* AST and ALT≤1.5 times the upper limit of normal (ULN);
* Total serum bilirubin≤1.5 times ULN;
* Hemoglobin≥90g/L;
* Platelet≥100000/ul;
* The creatinine in the normal range or creatinine clearance rate ≥60ml/min;
* Left ventricular ejection fraction (LVEF) ≥50%;
* Females of childbearing age are required to be practicing effective contraceptive measures and to have a negative serum or urine pregnancy test before study.
* Written informed consent is obtained.

Exclusion Criteria:

* included a history of or current brain metastases, clinically significant cardiovascular disease or uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 3 weeks
  Dose-limiting toxicity was defined as any one of the following (NCI-CTCAE Version 4.0): (a) hypertension: uncontrollable grade 3 hypertensive or grade 4. (b) reduced LVEF: 2 degrees or above. (c) neutropenia : 3 degrees or above. (d) thrombopenia: 3 degrees or above. (e) Other Non-hematologic toxicity (not including alopecia, nausea or vomiting): 3 degrees or above.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No